CLINICAL TRIAL: NCT06588907
Title: Evaluation of the Efficacy of Procedural Sedoanalgesia and Infraclavicular Nerve Blockade on Analgesia in Forearm Fractures in the Emergency Department
Brief Title: Pain Palliation in Forearm Fractures in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Sarcan, Doctor, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESarcan
Record Dates: First submitted 2024-07-08; First posted 2024-09-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Forearm Fracture; Radius Fractures; Ulnar Fracture
Keywords: Procedural sedation-analgesia; infraclavicular nerve block
MeSH Terms: conditions — Radius Fractures; Ulna Fractures | interventions — Bupivacaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): Reduction will be performed under procedural sedation analgesia (PSA)
  Interventions: Drug: Ketamine
- Group B (Active Comparator): Reduction will be performed under ultrasound-guided infraclavicular nerve block (ICB).
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — After preparing the infraclavicular block site, a 22-gauge needle, guided by ultrasound, will be placed in the 6-7 o'clock position in the same plane as the ultrasound probe. Subsequently, lateral, medial, and posterior cords described as hypoechoic nerve fascicles within hyperechoic structures will be identified. Initially, 2 mL of saline will be administered to confirm proper spread. Once confirmed, 20 mL of 0.25% bupivacaine (prepared by diluting 10 mL of 0.5% bupivacaine with 10 mL of normal saline) will be injected in fractional doses with intermittent negative aspiration. Fifteen minutes after this procedure, anesthesia depth will be assessed using a cold-hot test, followed by reduction and application of the cast.
  Other Names: Infraclavicular nerve block (ICB)
  Arms: Group B
Drug: Ketamine — Until the recovery period, patients will be closely monitored by an experienced doctor or nurse during sedation. Emergency equipment will be readily available in case of any complications. The following protocol will be used for procedural sedation-analgesia (PSA): Ketamine will be administered intravenously at a dose of 0.5-1 mg/kg. Patients with Numeric Rating Scale (NRS) scores above 5 may receive additional doses of 0.25-1 mg/kg, repeated every 5 to 10 minutes as needed.
  Other Names: procedural sedation-analgesia
  Arms: Group P

SUMMARY:
The aim is to evaluate the success of reduction procedures and pain palliation in patients with forearm fractures undergoing reduction under procedural sedation-analgesia (PSA) and ultrasound (US)-guided infraclavicular nerve block (ICB) in the emergency department.

DETAILED DESCRIPTION:
Forearm fractures are among the most frequent reasons for adults to visit the emergency department. These fractures cause significant pain both due to the fracture itself and during the reduction process. Pain management in emergency departments (ED) is crucial. Therefore, multimodal approaches are available to reduce or eliminate pain during the reduction process. The aim of this study is to evaluate the success and pain palliation of the reduction process with procedural sedation-analgesia (PSA) and with reduction under ultrasound (US)-guided infraclavicular nerve block (ICB) in patients with forearm fractures. The secondary aim is to compare patient comfort, physician comfort, side effects, length of stay in the emergency department, and the need for painkillers after discharge between these two procedures, and to identify the most suitable method. This study aims to contribute to practical applications in order to provide optimal pain control in patients with forearm fractures in emergency departments.

Patients' pain levels at arrival, pre-reduction procedure, and post-reduction procedure will be recorded using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain).The success of the reduction procedure, whether further reduction attempts were necessary, and findings from post-reduction control X-rays (radial height, radial tilt, and volar tilt) will be noted and evaluated by orthopedic physicians.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older,
* Diagnosed with forearm fracture using standard radiography,
* Hemodynamically stable individuals,
* Without vascular or nerve injury,
* Without infection in the skin or tissues where the needle will pass,
* Able to provide written and verbal consent and are capable of giving consent

Exclusion Criteria:

* Those with allergies to drugs used for sedoanalgesia and peripheral nerve blockade,
* Those who are hemodynamically unstable,
* Patients with ASA (American Society of Anesthesiologists) classification 3-4 will not be included in the group for whom PSA will be applied,
* Patients with coagulopathy, liver, or kidney failure,
* Patients with opioid, alcohol, or substance dependency,
* Those with skin infections or open wounds in the area where local anesthetic will be administered,
* Pregnant or suspected pregnant individuals,
* Those who do not provide written and verbal consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of patients' pain levels according to the Numerical Rating Scale (NRS) after the applied protocols. | 1. Pain level at the 1. minute upon presentation to the emergency room. 2. Pain level after the implementation of the protocols, i.e. 1 hour later. 3. Pain level 24 hours after the procedure.
  Pain levels at arrival, pre-reduction procedure, and post-reduction procedure will be recorded using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain).
Success of reduction following the applied protocols. | An x-ray will be taken before the reduction process, i.e. at 10 minutes. An x-ray will be taken at 1 hour after the reduction process.
  The success of the reduction procedure, whether further reduction attempts were necessary, and findings from post-reduction control X-rays (radial height, radial tilt, and volar tilt) will be noted and evaluated by orthopedic physicians.
Evaluation of the need for additional rescue treatments during the procedure. | Rescue analgesia will be administered if NRS is above 5 fifteen minutes after the protocols are applied.
  If NRS is above 5, as first-line rescue analgesia, tramadol 50 or 100 mg IV diluted in 100 mL normal saline will be administered over 15 minutes. If pain persists above NRS 5, second-line treatment with 50 mcg fentanyl diluted in 100 mL normal saline will be administered over 15 minutes.

SECONDARY OUTCOMES:
Patient and practitioner satisfaction with the reduction procedure. | The satisfaction survey for both the patient and the reduction practitioner will be conducted 30 minutes after the reduction procedure.
  Patient and reduction practitioner satisfaction will be recorded using a 5-point Likert scale (1: very poor, 2: poor, 3: neutral, 4: good, 5: very good).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Erdem, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

REFERENCES:
- [Background] Fauteux-Lamarre E, Burstein B, Cheng A, Bretholz A. Reduced Length of Stay and Adverse Events Using Bier Block for Forearm Fracture Reduction in the Pediatric Emergency Department. Pediatr Emerg Care. 2019 Jan;35(1):58-62. doi: 10.1097/PEC.0000000000000963. PMID 27918376
- [Result] Tekin E, Aydin ME, Turgut MC, Karagoz S, Ates I, Ahiskalioglu EO. Can ultrasound-guided infraclavicular block be an alternative option for forearm reduction in the emergency department? A prospective randomized study. Clin Exp Emerg Med. 2021 Dec;8(4):307-313. doi: 10.15441/ceem.20.136. Epub 2021 Dec 31. PMID 35000358
- [Result] Kukreja P, Kofskey AM, Ransom E, McKenzie C, Feinstein J, Hudson J, Kalagara H. Comparison of Supraclavicular Regional Nerve Block Versus Infraclavicular Regional Nerve Block in Distal Radial Open Reduction and Internal Fixation: A Retrospective Case Series. Cureus. 2022 Apr 12;14(4):e24079. doi: 10.7759/cureus.24079. eCollection 2022 Apr. PMID 35573547
- [Derived] Sarcan E, Erdem AB, Uysal SB, Duman E, Cebeci Z, Arik E. Pain management with ketamine procedural sedation and infraclavicular block for forearm fracture in the emergency department. Am J Emerg Med. 2025 Oct;96:256-263. doi: 10.1016/j.ajem.2025.07.012. Epub 2025 Jul 16. PMID 40694916

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT06588907/Prot_SAP_ICF_000.pdf